CLINICAL TRIAL: NCT03154177
Title: Group Antenatal/Postnatal Care in Rwanda: a Cluster Randomized Control Trial (RCT) to Measure Its Effectiveness on Increasing Gestational Age, Mortality Among Preterm and Low Birth Weight Infants
Brief Title: Group Antenatal/Postnatal Care in Rwanda
Acronym: PTBi Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Rwanda (Other); Rwanda Biomedical Centre (Other); Ministry of Health, Rwanda (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: A123218-Rw (UCSF RAS #)
Record Dates: First submitted 2017-04-14; First posted 2017-05-16 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pregnancy Complications; Preterm Birth; Preterm Labor; Stillbirth; Low Birth Weight; Neonatal Mortality
MeSH Terms: conditions — Pregnancy Complications; Premature Birth; Obstetric Labor, Premature; Stillbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard ANC and PNC care only (No Intervention): Standard care offered following national guidelines of ANC and PNC.
- Standard Care + Ultrasound+Pregnancy Testing (Other): Standard care in combination with early pregnancy testing and ultrasound.
  Interventions: Procedure: Ultrasound+Pregnancy Testing
- Group ANC and PNC only (Experimental): Health facilities randomized to provide group ANC/PNC.
  Interventions: Behavioral: Group ANC/PNC
- Group Care + Ultrasound+Pregnancy Testing (Experimental): Group ANC and PNC care, in combination with early pregnancy testing and ultrasound.
  Interventions: Behavioral: Group ANC/PNC; Procedure: Ultrasound+Pregnancy Testing

INTERVENTIONS:
Behavioral: Group ANC/PNC — The primary intervention is group antenatal and postnatal care wherein women receive their care in a group with other women with similar due dates. After an initial individual visit all care is given in groups although the majority of the time is dedicated to facilitated discussion and women can come for additional acute care if needed. Group antenatal care will be three group visits between 20 and 40 weeks gestation and group postnatal care will be one group visit and approximately 6 weeks post delivery.
  Arms: Group ANC and PNC only; Group Care + Ultrasound+Pregnancy Testing
Procedure: Ultrasound+Pregnancy Testing — Half of all study sites will receive early pregnancy testing, conducted by community health workers at community level and ultrasound for gestational age dating and early screening at the health center.
  The primary analysis will not assess the effectiveness of this intervention.
  Arms: Group Care + Ultrasound+Pregnancy Testing; Standard Care + Ultrasound+Pregnancy Testing

SUMMARY:
The focus of this work is to improve antenatal care (ANC) and postnatal care (PNC) at the health center level in five districts in Rwanda (Bugesera, Burera, Nyamasheke, Nyarugenge, and Rubavu). 36 health centers in these districts are included in this cluster randomized control trial (RCT) of group ANC and PNC care to measure this alternative model's effects on gestational age at birth, survival of preterm and low birth weight infants at 42 days of life, and ANC and PNC coverage. To improve antenatal assessment of gestational age, nurses will be trained in obstetric ultrasound at 18 health centers. These facilities will also incorporate pregnancy testing with urine dipstick to be performed by community health workers in charge of maternal health to facilitate early entry into ANC. This trial will test the hypothesis that women who participate in this alternative model of group ANC will experience increased gestational age at birth, as compared to women who receive standard focused ANC. This study is a collaboration with the University of Rwanda, the Rwandan Ministry of Health (MOH), the Rwanda Biomedical Center, and UCSF.

The group care model used in this study is Rwanda-specific model developed by a Rwandan technical working group. The model includes an individual clinical visit for the first antenatal visit, followed by three group visits spaced about 8 weeks apart throughout pregnancy and a postnatal group visit at approximately 6 weeks after birth. Women will be grouped into stable groups of approximately 8-12 women with similar due dates. A community health worker (CHW) and a health center nurse will work together as co-facilitators to lead each of the groups. Each group visit includes clinical assessment, education, and treatments as appropriate for the women who attend. The model is founded on facilitative leadership of the groups, in which the co-facilitators allow women's experiences and interests to drive the content and women are encouraged to help one another cope with obstacles to optimal health. Facilitators will be supported by master trainers who will visit health centers to observe group sessions and offer supportive feedback.

Data collected in this trial will include measures of the satisfaction of both women and providers with the group care, content of care differences between standard and group care, and perinatal outcomes such as gestational age at delivery and 42-day preterm and low birth weight infant survival.

DETAILED DESCRIPTION:
This study aims to determine the effect of a group care model, which incorporates both group care antenatal (ANC) and postnatal care (PNC), on the following:

1. Gestational age (GA) at birth;
2. Adherence to the recommended four ANC and one facility-based PNC visits; and
3. Mortality at 42 days among preterm and low birth weight infants.

In this cluster RCT at the health center level, facilities will be pair-matched based on factors affecting GA at delivery such as monthly ANC enrollment, quality of ANC and PNC delivery, potential lost-to-follow-up (LTFU) rate, and additional criteria pertaining to facility capacity. Within each pair, a facility will be randomly chosen to implement the intervention, group ANC and PNC, while the control facility will continue to provide standard ANC and PNC. Pairs will then be further matched with other pairs into quadruples (to the extent possible), within which one pair will be assigned to additionally implement ultrasound at the health center level and early pregnancy testing at the community level. Overall, each facility will have one of the following assignments:

* Arm 1: Standard ANC and PNC care only
* Arm 2: Standard ANC and PNC care, with the addition of early pregnancy testing and ultrasound
* Arm 3: Group ANC and PNC only
* Arm 4: Group ANC and PNC care, with the addition of early pregnancy testing and ultrasound

This design will allow a primary analysis on the difference between group care and standard care and will also make it possible to assess the effect of early pregnancy testing in the community and obstetric ultrasound at the health center on early entry into ANC and number of visits attended.

The Rwanda group ANC/PNC model was developed by a Technical Working Group of representatives from maternal-child health stakeholders in Rwanda. Key characteristics:

1. Women sit in a circle in a group space where confidentiality and mutual respect are prioritized. Key messages consistent with Rwanda's ANC/PNC packages are delivered through facilitated discussion; women speak more than the facilitators.
2. Women and newborns receive the routine assessments, screening, and treatments described in the Rwanda guidelines, as well as treatments indicated for special conditions. Health assessments are conducted at the start of the visit, and women participate as much as possible in their own self-assessments. Individual consultations with facilitators are conducted in a semi-private area.
3. Two co-facilitators lead each group visit (one midwife/nurse and one CHW). Co-facilitators "debrief" after every group visit in a continuous learning and quality improvement process. The group care co-facilitators are trained and supported by 6 Rwandan Master Trainers.
4. Women can return to the health facility at any time for evaluation of danger signs or other concerns. Referrals to the district hospital are done per current national guidelines.

Both control and intervention sites, as well as district hospitals that may receive referrals from our study sites, will receive the initial intervention of data strengthening and training around data use activities so as to improve the quality of data being collected and strengthen outcome measurement within all facilities involved in the study

Additionally, in order to evaluate other secondary outcomes, data will also be collected through: (1) questionnaires administered to a random sample of ANC and PNC participants and all providers at baseline and different time points throughout the study; (2) observations and debriefs of group care sessions; (3) qualitative research around acceptability of the group model from participants and providers; (4) cost-effectiveness analysis of the group care model.

ELIGIBILITY:
Individual inclusion Criteria:

Women receiving ANC and PNC care

* all women who enroll in ANC -including pregnant adolescents
* primary data analysis will be restricted to those women in the intervention and control facilities who present for ANC 1 before 24 weeks gestation and have attended more than 1 ANC visit at the health facility.

Providers • Currently provide antenatal or postnatal care

Individual exclusion Criteria:

Women receiving ANC and PNC care

* women who present for ANC 1 after 24 weeks gestation
* women who do not attend more than 1 ANC at the health facility will be excluded from the primary analysis

Providers

• Providers that do not provide antenatal or postnatal care

Site-level exclusion criteria:

• sites that have less than 2 ANC providers.

Site-level inclusion criteria:

• Study sites that have at least 2 ANC providers were included in the final selection of 36 sites. The following are study sites by district:

Nyamasheke District Nyamasheke Kibingo Mugera Mwezi Karengera Kibogora Gisakura Yove

Nyarugenge District Cor-unum Biryogo Rugarama Kabusunzu

Rubavu District Murara Nyakiriba Busasamana Karambo Gisenyi Kigufi Mudende

Bugesera District Ruhuha Gakurazo Gashora Ngeruka Kamabuye Nyamata Ntarama Juru Mayange Nzangwa Nyarugenge

Burera District Cyanika Kirambo Ndongozi Gitare Gahunga Mucaca

Ages: 13 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only female participants are being studied (assuming mom's will be source of GA measurement at delivery).
Enrollment: 26381 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Gestational Age | within the first 3 days after delivery
  Average gestational age at delivery among women who enroll in ANC before 24 weeks of gestation and had at least 2 ANC visits at that facility.

SECONDARY OUTCOMES:
Preterm birth rate | At delivery
  Proportion of preterm deliveries among mothers enrolled in ANC
Preterm 28-day and 42-day mortality rate | 28 days and 42 days post delivery
  28-day and 42-day mortality rate among preterm infants whose mother enrolled in ANC
Women who adhered to four ANC visits | From the day of first ANC visit at the health center until the day of delivery
  Proportion of women who adhered to four ANC visits among all mothers who have received at least one ANC visit at facility.
Adherence to 6 week postnatal visit | 42 days post delivery
  Proportion of women who adhered to the 6-week PNC visit at the health center among those who attended at least 2 ANC at the facility.
1st ANC visit during the first trimester | up to 14 weeks gestation
  Proportion of women with 1st ANC visit during the first trimester among those who have at least one ANC visit.
High-risk Women | From the day of first ANC visit at the health center until the day of delivery
  Proportion of women identified during ANC as being high-risk
C-section deliveries | At Delivery
  Proportion of pregnancies resulting in C-section deliveries among those enrolled in ANC at facility.
Newborns with neonatal morbidities, specifically, jaundice, rapid breathing, fever, pneumonia, hypothermia, and/or cord infection | 28 days post delivery
  Proportion of newborns with neonatal morbidities, specifically, jaundice, rapid breathing, fever, pneumonia, hypothermia, and/or cord infection, among all those whose mother received ANC at facility, and among all those who received PNC at facility.

OTHER OUTCOMES:
Cost-effectiveness | Costs will be measured prospectively from baseline through the end of the intervention once sample size is achieve--approximately 18 months from baseline.
  Costs of ANC delivery and program costs will be collected prospectively, and costs associated with each adverse outcome that may be potentially averted will be calculated. Effectiveness measures will be: number of deliveries conducted by skilled health workers; total number of ANC visits, first ANC visit before 16 weeks and 4 standard ANC visits completed; and number of preterm births prevented.
Qualitative assessment of group care feasibility and acceptability to women and providers | up to 18 months
  Qualitative work (in-depth interviews and focus group discussions) with women and providers to inform any fine tuning to the model will be conducted at 9 and 18 months after implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Dilys Walker, MD, Principal Investigator — University of California, San Francisco; Sabine F Musange, MD, MSc, Principal Investigator — University of Rwanda
Locations (2):
- Rwanda (2):
  - Rwanda Biomedical Center, Kigali
  - University of Rwanda, Kigali

IPD SHARING:
Plan to Share IPD: Undecided
Data from the study will be shared, but the extent to which individual participant data can be shared is yet to be determined. This will be done to the extent possible, conforming to any partner requirements or Rwanda IRB requirements.

REFERENCES:
- [Background] Lincetto O, Mothebesoane-Anoh S, Gomez P, Munjanja S. Antenatal care. Chapter 2. Opportunities for Africa's Newborns.
- [Background] Bhutta ZA, Das JK, Bahl R, Lawn JE, Salam RA, Paul VK, Sankar MJ, Blencowe H, Rizvi A, Chou VB, Walker N; Lancet Newborn Interventions Review Group; Lancet Every Newborn Study Group. Can available interventions end preventable deaths in mothers, newborn babies, and stillbirths, and at what cost? Lancet. 2014 Jul 26;384(9940):347-70. doi: 10.1016/S0140-6736(14)60792-3. Epub 2014 May 19. PMID 24853604
- [Background] National Institute of Statistics of Rwanda. (2015). Demographic and Health Survey 2014-2015: Key Findings.
- [Background] Ickovics JR, Kershaw TS, Westdahl C, Magriples U, Massey Z, Reynolds H, Rising SS. Group prenatal care and perinatal outcomes: a randomized controlled trial. Obstet Gynecol. 2007 Aug;110(2 Pt 1):330-9. doi: 10.1097/01.AOG.0000275284.24298.23. PMID 17666608
- [Background] Catling CJ, Medley N, Foureur M, Ryan C, Leap N, Teate A, Homer CS. Group versus conventional antenatal care for women. Cochrane Database Syst Rev. 2015 Feb 4;2015(2):CD007622. doi: 10.1002/14651858.CD007622.pub3. PMID 25922865
- [Background] Maternal Health Task Force, Harvard School of Public Health, et al. Group Care. Innovative Methods 2014.
- [Background] Prost A, Colbourn T, Seward N, Azad K, Coomarasamy A, Copas A, Houweling TA, Fottrell E, Kuddus A, Lewycka S, MacArthur C, Manandhar D, Morrison J, Mwansambo C, Nair N, Nambiar B, Osrin D, Pagel C, Phiri T, Pulkki-Brannstrom AM, Rosato M, Skordis-Worrall J, Saville N, More NS, Shrestha B, Tripathy P, Wilson A, Costello A. Women's groups practising participatory learning and action to improve maternal and newborn health in low-resource settings: a systematic review and meta-analysis. Lancet. 2013 May 18;381(9879):1736-46. doi: 10.1016/S0140-6736(13)60685-6. PMID 23683640
- [Derived] Sayinzoga F, Lundeen T, Musange SF, Butrick E, Nzeyimana D, Murindahabi N, Azman-Firdaus H, Sloan NL, Benitez A, Phillips B, Ghosh R, Walker D. Assessing the impact of group antenatal care on gestational length in Rwanda: A cluster-randomized trial. PLoS One. 2021 Feb 2;16(2):e0246442. doi: 10.1371/journal.pone.0246442. eCollection 2021. PMID 33529256
- [Derived] Musange SF, Butrick E, Lundeen T, Santos N, Azman Firdaus H, Benitez A, Nzeyimana D, Kayiramirwa Murindahabi N, Nyiraneza L, Sayinzoga F, Ndahindwa V, Ngabo F, Condo J, Walker D. Group antenatal care versus standard antenatal care and effect on mean gestational age at birth in Rwanda: protocol for a cluster randomized controlled trial. Gates Open Res. 2019 Sep 27;3:1548. doi: 10.12688/gatesopenres.13053.1. eCollection 2019. PMID 31656954
- [Derived] Lundeen T, Musange S, Azman H, Nzeyimana D, Murindahabi N, Butrick E, Walker D. Nurses' and midwives' experiences of providing group antenatal and postnatal care at 18 health centers in Rwanda: A mixed methods study. PLoS One. 2019 Jul 11;14(7):e0219471. doi: 10.1371/journal.pone.0219471. eCollection 2019. PMID 31295335
- [Derived] Musabyimana A, Lundeen T, Butrick E, Sayinzoga F, Rwabufigiri BN, Walker D, Musange SF. Before and after implementation of group antenatal care in Rwanda: a qualitative study of women's experiences. Reprod Health. 2019 Jun 27;16(1):90. doi: 10.1186/s12978-019-0750-5. PMID 31248425